CLINICAL TRIAL: NCT02162186
Title: Analysis of Clinical Outcome and Implant Migration of the Cementless Tri-Fit Total Hip Replacement System
Brief Title: Clinical and Radiographic Outcomes of the Corin Tri-Fit Total Hip Replacement
Status: Completed | Type: Observational
Sponsor: Corin (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP2013-12
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2018-11

CONDITIONS: Osteoarthritis of Hip; Congenital Hip Dysplasia; Avascular Necrosis
Keywords: Arthroplasty, Replacement, Hip/methods; Hip Joint/physiopathology; Hip Joint/radiography; Hip Joint/surgery; Hip Prosthesis; Outcome Assessment (Health Care); Female; Male; Adult
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Dislocation, Congenital; Osteonecrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The study will evaluate the radiographs (x-rays) of 100 patients with a TriFIT total hip at 2 weeks, 3 months, 6 months, 12 months, and yearly following surgery to see if there has been any movement or wear in the hip stem over the course of the study. The study will also record clinical data on each patient using various functional tests and questionnaires at the same intervals.

DETAILED DESCRIPTION:
The present study will prospectively recruit 100 patients scheduled for elective total hip replacement with Corin's TriFIT Hip System at the Ottawa Hospital - General Campus. As part of their clinical care, patients routinely undergo a clinical examination and have had radiographs taken at 2 weeks, 3 months, 6 months, 12 months, and yearly following surgery. Using specialized software, radiographs from each interval will be examined to assess femoral stem migration and joint wear patterns. Femoral stem migration will be assessed using computer-assisted software. The study will also assess the rate of implant failure during the first two post-operative years. Clinical assessments and questionnaires will also be completed during each of the follow-up intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for primary, unilateral total hip replacement (THR) with no previous history of hip replacement and/or fracture surgery.
* Patients with arthritis secondary Noninflammatory Degenerative Joint Diseases (NIDJD), including osteo/degenerative arthritis, congenital hip dysplasia, and avascular necrosis.
* Patients who do not meet any of the exclusion criteria.

Exclusion Criteria:

* Patients with previous fusions, acute femoral neck fractures, above knee amputations, or previous total knee replacement.
* Patients who had previously undergone an ipsilateral hemi resurfacing, total resurfacing, total bipolar, unipolar or total hip replacement device.
* Patients with neuropathic joints.
* Patients who required structural bone grafts.
* Patients with an ipsilateral girdlestone.
* Patients who otherwise met the study criteria, but for which appropriate clinical follow-up data is not available (i.e. patients deceased prior to 2-year follow-up, patients refused to return for follow-up).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The first 100 patients Dr. Paul Beaule undergoing a total hip replacement with Corin's TriFIT Total Hip replacement system that meet the eligibility requirements and consent to do the study.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2014-10; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Femoral Stem Migration Radiographic Assessment | 2 weeks to end of study (approximately 2 years) post-operatively
  Femoral stem migration (in millimeters (mm)) will be assessed using computer-assisted Einzel Bild Roentgen Analyze-Femoral Component Analysis (EBRA-FCA) software and radiographs taken at each interval.
Rate of Implant Failure | 2 weeks to end of study (approximately 2 years) post-operatively
  The number of revisions will be recorded.
Radiographic Assessment of Wear in the Acetabular Components | 2 weeks to end of study (approximately 2 years) post-operatively
  Anterior-posterior (AP) and lateral radiographs from each follow-up visit will be used to assess wear of the acetabular (hip) components.

SECONDARY OUTCOMES:
Harris Hip Score (HHS) | 2 weeks to end of study (approximately 2 years) post-operatively
  A standardized set of questions and measurements to assess the function of the hip. It includes pain, function, range of motion (ROM), and absence of deformity.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 2 weeks to end of study (approximately 2 years) post-operatively
  A standardized set of questions and measurements to assess the function of the hip. It includes pain, stiffness, and joint function.
SF (Short Form)-12 Questionnaire | 2 weeks to end of study (approximately 2 years) post-operatively
  A subject-completed questionnaire with questions and he/she's health and well-being.
UCLA (University of California, Los Angeles) Activity Level | 2 weeks to end of study (approximately 2 years) post-operatively
  A subject-completed questionnaire which asks his/her current activity level.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Beaule, MD, Principal Investigator — Ottawa Hospital
Locations (1):
- Ottawa Hospital - General Campus, Ottawa, Ontario, Canada